CLINICAL TRIAL: NCT07274228
Title: Risk of Serious Adverse Events Associated With Tamsulosin Use in Older Adults With Advanced Chronic Kidney Disease: A Population-Based Cohort Study Research Protocol
Brief Title: Tamsulosin and the Risk of Serious Adverse Events
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 2025 0906 600 000; ICES # 2025 0906 600 000 (Other: ICES, Ontario, Canada)
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: Chronic kidney disease; High-throughput computing; Tamsulosin; Adverse events; Older adults; Cohort study; Drug safety
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Tamsulosin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low dose of tamsulosin (0.4 mg/day (standard dose)): Residents of Ontario, male, aged 66 years or older with advanced CKD (an eGFR <45 mL/min per 1.73 m² but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for tamsulosin (low dose 0.4 mg/day) at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 01, 2008, to December 01, 2024. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, with each patient entering the cohort only once. If the investigators conduct the study in Alberta, the accrual period for Alberta will be determined.
  Interventions: Drug: Tamsulosin
- High dose of tamsulosin (0.8 mg/day (off label dose)): Residents of Ontario, male, aged 66 years or older with advanced CKD (an eGFR <45 mL/min per 1.73 m² but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for tamsulosin (high dose 0.8 mg/day) at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 01, 2008, to December 01, 2024. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, with each patient entering the cohort only once. If the investigators conduct the study in Alberta, the accrual period for Alberta will be determined.
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin — The primary exposure of interest will be oral tamsulosin at a dose of 0.4 mg/day, representing the median dose in high-throughput computing analyses. For the primary comparison, oral tamsulosin at a dose of 0.4 mg/day will be chosen to reduce the influence of indication bias.
  Other Names: APO-Tamsulosin CR; AURO-Tamsulosin CR; Flomax CR [DSC]; JAMP-Tamsulosin; RATIO-Tamsulosin [DSC]; SANDOZ Tamsulosin; SANDOZ Tamsulosin CR; TEVA-Tamsulosin CR; TEVA-Tamsulosin [DSC]

SUMMARY:
This is a population-based cohort study assessing whether initiating a higher dose of tamsulosin (0.8 mg/day) compared to a lower dose (0.4 mg/day) in older adults with advanced chronic kidney disease (CKD) (an estimated glomerular filtration rate (eGFR) <45 mL/min per 1.73 m² but not receiving dialysis or having a history of kidney transplantation) is associated with a higher 90-day risk of a composite outcome of all-cause hospitalization or all-cause emergency visits or all-cause mortality.

DETAILED DESCRIPTION:
*Summary*

Background:

Tamsulosin, an alpha-1a adrenergic receptor blocker, primarily used to treat benign prostate hyperplasia (BPH). Despite its significant renal elimination, there are no clear safety guidelines for its use in patients with CKD, raising important safety concerns. Using a novel high-throughput approach using Ontario healthcare databases, the investigators identified an increased risk of adverse outcomes in patients with advanced CKD (an eGFR <45 mL/min/1.73 m² but not receiving dialysis or having a history of kidney transplantation) who were newly prescribed tamsulosin compared to a similar cohort of non-users.

To validate these findings, the investigators plan to conduct a population-based cohort study among older adults in Ontario, Canada, comparing the risk of serious adverse events among those initiating a higher dose versus a lower dose of tamsulosin in the outpatient setting.

Methods: The study will include older adults (≥ 66 years) with eGFR <45 mL/min/1.73 m² (not receiving dialysis or having a history of kidney transplantation) who were dispensed a new outpatient prescription for oral tamsulosin. In Ontario, the sample will be accrued from January 1, 2008, through December 01, 2024. The prescription date will be the index date (start of cohort follow-up). Older adults initiating treatment with tamsulosin will be divided into two groups based on their dosage: high dose (0.8 mg/day, off-label) and low dose (0.4 mg/day, standard dose). Propensity score weighting will be used to ensure both groups are well-balanced on a comprehensive set of measured baseline characteristics.

The Patient outcome will be a 90-day composite of all-cause hospitalization, emergency department visit, or mortality.

*Background*

Tamsulosin, a selective alpha-1 adrenergic receptor antagonist widely used for BPH, is frequently prescribed to older adults, including those with CKD, despite limited safety data in this population.

Tamsulosin is primarily eliminated through the kidneys, with approximately 76% excreted unchanged. Pharmacokinetic studies on tamsulosin demonstrated that low eGFR alters the pharmacokinetics of tamsulosin primarily through changes in protein binding rather than reduced renal excretion. In patients with low eGFR, increased levels of alpha-1-acid glycoprotein (a1-AGP) led to higher total plasma concentrations, but unbound (active) tamsulosin levels remained stable, suggesting minimal impact on pharmacologic effects. Current prescribing guidelines from UpToDate and product monograph, recommended no dosage adjustment for tamsulosin in patients with creatinine clearance (CrCl) ≥10 mL/min. However, for patients with severe CKD (CrCl <10 mL/min) or those on hemodialysis, tamsulosin pharmacokinetics have not been thoroughly studied. Given its high protein binding and minimal renal excretion of the active (unbound) form, dose adjustments may not be necessary, but caution is advised due to increased total plasma concentrations and potential for adverse effects, particularly hypotension, dizziness, syncope. According to the product monograph, though rare, some serious and potentially fatal side effects of tamsulosin include severe dizziness, falls, fractures, ejaculation issues, and prolonged or painful erections. Case reports and trials also highlight other adverse events like severe hypotension, cardiovascular events, and delirium. Notably, there are no clear guidelines addressing the safety of tamsulosin in patients with CKD.

Using a high-throughput drug-safety computing approach, investigators previously identified a potential 30-day increased risk of emergency visits, hospitalizations, and mortality after initiating tamsulosin. Understanding the risks of initiating higher versus lower doses of tamsulosin in older adults with low kidney function can be used to guide safe prescribing and better outcomes in this population.

*Objectives*

Is there a higher 90-day risk of a composite outcome of all-cause hospitalizations or all-cause emergency visits or all-cause mortality among older adults with advanced CKD (an eGFR <45 mL/min per 1.73 m² but not receiving dialysis or having a history of kidney transplantation) who initiate a higher dose (off-label dose: 0.8 mg/day) vs lower dose (standard dose: 0.4 mg/day) of tamsulosin in the outpatient setting?

*Study Design and Setting*

The investigators propose a population-based retrospective cohort study using linked administrative health data from Ontario, Canada. If the Ontario cohort is small to generate reliable estimates, the investigators will augment the study by performing an analysis using Alberta health administrative data.

Ontario data will be sourced from ICES (ices.on.ca). It offers secure, encrypted individual-level data for Ontario residents, all with universal access to hospital and physician services under a government-funded, single-payer healthcare system. The use of data in this study is authorized under section 45 of Ontario's Personal Health Information Protection Act, which does not require review by a research ethics board. The information needed for analyzing the primary outcomes is available across specific databases within the ICES system: data on all-cause hospitalizations are available in the Canadian Institute for Health Information Discharge Abstract Database, emergency visits in the National Ambulatory Care Reporting System, and mortality in the Registered Persons Database.

If the investigators proceed with conducting the study in Alberta, the Alberta data will be accessed through the Alberta Kidney Disease Network (AKDN). This dataset ends in ~ 2021.

The investigators are publicly registering our study protocol and documenting the study description, design, and statistical analysis prior to conducting outcome analyses. The results of this study will be reported adhering to RECORD reporting guidelines.

*Study Population*

The investigators will include all older men (≥66 years) with an eGFR <45 mL/min per 1.73 m² (not receiving dialysis or having a history of kidney transplantation) who received a new outpatient prescription for oral tamsulosin at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 1, 2008, to December 01, 2024. The dispensing date of the prescription will serve as the index date, and only the first eligible prescription will be included to ensure unique cohort entry, and each individual can enter the cohort only once.

*Baseline Characteristics*

Health records, census files, hospital discharge records, laboratory data, and physician claims will provide baseline variables, including demographic characteristics (such as age, sex, rurality, neighborhood income quintile), comorbidities, and medication use. Baseline comorbidities and healthcare utilization will be assessed using 5-year and 1-year look-back periods from the index date. Baseline medication use will be assessed within 120 days prior to the index date.

*Statistical analysis plan*

Software:

All statistical analyses will be conducted using SAS software version 9.4 (SAS Institute, Cary, NC).

Descriptive Statistics:

Categorical variables will be reported as frequencies and proportions, while continuous variables will be presented as means with standard deviations (SD) or medians with interquartile ranges (IQR), as appropriate. Differences in baseline characteristics between the high-dose (0.8 mg/day, off-label) and low dose (0.4 mg/day, standard dose) groups will be examined using standardized differences, with differences ≥10% considered meaningful.

Balancing comparator group:

The investigators will use the inverse probability of treatment weighting on the propensity score to balance baseline characteristics between the high dose and low dose groups based on their baseline characteristics, including known indicators for tamsulosin use.

The investigators will conduct multivariable logistic regression analyses to generate propensity scores using all baseline characteristics. Average treatment effect in the treated (ATT) weights will be used, where patients in the low dose group will be assigned weights calculated as (propensity score / [1 - propensity score]). In contrast, patients in the high dose group will receive a weight of 1. This method will produce a weighted pseudo sample of patients in the referent group (i.e. low-dose: tamsulosin 0.4 mg/day, standard dose) with a similar distribution of measured characteristics as the high-dose (tamsulosin 0.8 mg/day, off-label) group. Baseline characteristics between groups will be compared using standardized differences in unweighted and weighted samples, with differences exceeding 10% considered meaningful.

Regression analysis:

To evaluate the primary outcome composite measure of all-cause hospitalization or all-cause emergency department visits or all-cause mortality-the investigators will apply a modified Poisson regression analysis to estimate the risk ratio (RR) with 95% confidence intervals (CIs) and a binomial regression to estimate the risk difference (RD) with 95% CIs using the weighted cohort, with low-dose tamsulosin (0.4mg/day) group as the referent.

Secondary analysis:

The investigators will conduct independent testing for all secondary and mechanistic outcomes without adjusting for multiple comparisons. Each test will be performed and reported independently. In line with the best practices, the investigators will present the P-value for the primary outcome and report all secondary and mechanistic outcomes using point estimates with 95% confidence intervals, acknowledging them as exploratory analyses.

Additional analysis:

The investigators will conduct four additional analyses.

1. Effect measure modification (EMM):

   For EMM, the investigators will expand our cohort to all the eGFR levels and categorize them into three groups: eGFR ≥60, 45-<60, and <45 mL/min/1.73 m². Baseline characteristics between high-dose (0.8 mg/day) and low-dose (0.4 mg/day) tamsulosin groups will be assessed using standardized differences for all renal function categories combined and then within each of three eGFR categories (≥60, 45-<60, and <45 mL/min/1.73 m²).

   To further balance baseline characteristics between high-dose and low-dose tamsulosin groups, the investigators will apply the IPTW method (described above), based on propensity scores for all the eGFR categories combined and within each of the three eGFR categories.

   EMM will be assessed on both the additive and multiplicative scales.
   * For additive interaction, the investigators will use binomial regression with an identity link to estimate risk differences, including an interaction term between low-dose and high-dose tamsulosin groups and eGFR strata.
   * For multiplicative interaction, the investigators will use modified Poisson regression analysis to estimate risk ratios, including an interaction term between low-dose and high-dose tamsulosin groups and eGFR strata.
2. The investigators will conduct a pre-specified subgroup analysis of the primary outcome stratified by pre-2020 (which overlaps with high-throughput computing) (January 1, 2008, to March 01, 2020) and post-2020 (which does not overlap with high-throughput computing) (March 02, 2020, to December 01, 2024). The investigators will examine whether the association between higher-dose vs. lower-dose tamsulosin and the primary outcome is different (modified) in 2 period categories (the period prior to the end date of the high-throughput computing, and the period after the end-date of the high-throughput computing).
3. In a cohort of new users of tamsulosin, the investigators will compare the risk of toxicity between those who initiate a higher dose (off-label dose: 0.8 mg/day) and those on a lower dose (standard dose: 0.4 mg/day) of tamsulosin in the outpatient setting, versus non-users, specifically in older adult patients with advanced CKD (eGFR <45 mL/min per 1.73 m²). The investigators will apply the primary study outcomes, utilize the same baseline characteristics, and employ the statistical analysis methods used in the primary analysis.
4. The investigators will perform E-value analyses to determine the minimum association strength an unmeasured confounder would need with both the prescription drug and the outcome of interest (while adjusting for measured covariates) to eliminate the observed association.

*Combining Outcome Results from Ontario and Alberta*

This approach will only be used if the investigators proceed with conducting the analysis in Alberta.

Privacy preserving methods:

The investigators plan to use a privacy-preserving Cox-based approach for estimating risk ratios for multisite studies where individual-level data cannot be shared due to privacy constraints described by Shu et al. (2025). The proposed method requires only a single transfer of summary-level outputs from each province to the research team. It produces results identical to those from a corresponding log-binomial regression with combined individual-level data. The method was developed by adapting the risk-set table approach for survival outcomes, assuming stratified province-specific baseline risks, and allowing for confounding mitigation strategies such as propensity score matching or weighting to be done individually in each province. Each province will independently calculate these summary tables using their individual-level data. The summary-level risk-set tables generated in Alberta will be shared in a single data transfer to the coordinating site's analyst where they will be used to estimate the combined risk ratios and 95% confidence intervals. This will enable a robust and consistent analysis while maintaining data privacy and adhering to regulatory compliance. To comply with privacy regulations for minimizing the chance of identification of any individual, in all manuscripts, numbers of individuals are suppressed in the case of 5 or fewer participants (reported as ≤5). All team members will sign any required data confidentiality and data use agreements.

ELIGIBILITY:
Inclusion Criteria:

The cohort will include older adult men aged 66 years or older with advanced CKD (an eGFR <45 mL/min per 1.73 m² but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for tamsulosin at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 1, 2008, to December 01, 2024. The age criterion is set to guarantee that individuals in this population had at least one year of prior prescription drug coverage. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, with each patient entering the cohort only once.

Exclusion Criteria:

1. Data cleaning exclusions (e.g., individuals with missing or invalid age or administrative database number, OHIP ineligible on index date, death on or before the index date, non-Ontario residents). The investigators anticipate that very few records will be excluded due to data cleaning.
2. The investigators will exclude patients receiving tamsulosin doses other than 0.4mg/day or 0.8mg/day.
3. To ensure that patients are new tamsulosin users, the investigators will exclude those with any evidence of tamsulosin use in the 180 days before the index date.
4. Patients with more than one study drug prescription on the index date will be excluded, as this complicates the ability to ascertain the prescribed dose accurately.
5. The investigators will exclude patients with a prescription of Alpha1 blocker (alfuzosin, doxazosin, prazosin, silodosin, terazosin), 5 Alpha Reductase inhibitor (dutasteride, finasteride, dutasteride & tamsulosin), and non-oral study drugs in the previous 180 days, including the index date.
6. Individuals with end-stage renal disease, chronic dialysis, or a kidney transplant prior to the index date.
7. Evidence with hospital discharge or emergency department visit in the two days prior to or on the index date to ensure a new outpatient prescription.
8. Patients with no outpatient serum creatinine measurement 0- 365 days before the index date will be excluded.
9. Patients with unstable baseline kidney function (If the most recent serum creatinine test before the index date was an inpatient test [ER or hospitalization] <refer to this as test date 1>, and there is not at least one 'outpatient' serum creatinine in the year before test date 1) (If the most recent prior serum creatinine test before the index date was an inpatient test [ER or hospitalization] <refer to this as tests test date 1>, and while there is at least 'outpatient' serum creatinine test in the year before <test date 1>, the most recent outpatient test before <test date 1> differs by an eGFR 10 mL/min/1.73 m2 or more from the value on <test date 1>) will be excluded. In Ontario, it has been shown that outpatient serum creatinine measurements in the province, conducted on a single occasion, indicate stable values.
10. If more than one eligible prescription is available, restrict it to the first. The date of this prescription will be the index date

Min Age: 66 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Men aged 66 years or older with advanced CKD (eGFR <45 mL/min per 1.73 m² but not receiving dialysis or having a history of kidney transplantation) who have filled at least one outpatient prescription for oral tamsulosin between 2008 and 2024 in Ontario.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with a composite outcome of all-cause hospitalization or all-cause emergency visits, or all-cause mortality | Exposed cohort to tamsulosin (high dose (0.8 mg/day) versus low dose (0.4 mg/day) will enter the cohort and will be followed until study outcome (first event), death, or 90 days from the cohort entry date.
  All-cause hospitalization, all-cause emergency visits, and all-cause mortality will be combined into a composite measure. Only the first hospitalization or first emergency department visit occurring within 90 days after the cohort entry date will be considered.

SECONDARY OUTCOMES:
Number of participants with all-cause hospitalization | Exposed cohort to tamsulosin (high dose (0.8 mg/day) versus low dose (0.4 mg/day) will enter the cohort and will be followed until study outcome (first event), death, or 90 days from the cohort entry date.
  One of the components of the primary composite outcome, all-cause hospitalization, individually presented as a secondary outcome. Only the first hospitalization occurring within 90 days after the cohort entry date will be considered.
Number of participants with all-cause emergency department visits | Exposed cohort to tamsulosin (high dose (0.8 mg/day) versus low dose (0.4 mg/day) will enter the cohort and will be followed until study outcome (first event), death, or 90 days from the cohort entry date.
  One of the components of the primary composite outcome, all-cause emergency department visit, individually presented as a secondary outcome. Only the first emergency department visit occurring within 90 days after the cohort entry date will be considered.
Number of participants with all-cause mortality | Exposed cohort to tamsulosin (high dose (0.8 mg/day) versus low dose (0.4 mg/day) will enter the cohort and will be followed until study outcome (first event), death, or 90 days from the cohort entry date.
  One of the components of the primary composite outcome, all-cause mortality, individually presented as a secondary outcome.

OTHER OUTCOMES:
90-day composite outcome of a hospital encounter with atrial fibrillation/flutter or other arrhythmia | Exposed cohort to tamsulosin (high dose (0.8 mg/day) versus low dose (0.4 mg/day) will enter the cohort and will be followed until study outcome (first event), death, or 90 days from the cohort entry date.
  90-day hospital encounter (hospital admission or emergency visit) composite of atrial fibrillation/flutter or other arrhythmia (including pacemaker insertion, palpitations, tachycardia unspecified, atrioventricular block, supraventricular tachycardia, other conduction disorders, implantable cardiac defibrillator)
90-day composite outcome of a hospital encounter with heart failure or myocardial infarction, or ischemic stroke | Exposed cohort to tamsulosin (high dose (0.8 mg/day) versus low dose (0.4 mg/day) will enter the cohort and will be followed until study outcome (first event), death, or 90 days from the cohort entry date.
  90-day hospital encounter (hospital admission or emergency visit) with composite outcome of heart failure or myocardial infarction (most responsible diagnosis), or ischemic stroke (most responsible diagnosis)
90-day composite outcome of a hospital encounter with falls, hypotension, syncope, or hospital admission with receipt of an urgent computed tomography scan of the head | Exposed cohort to tamsulosin (high dose (0.8 mg/day) versus low dose (0.4 mg/day) will enter the cohort and will be followed until study outcome (first event), death, or 90 days from the cohort entry date.
  90-day hospital encounter (hospital admission or emergency visit) with composite outcome of falls, hypotension, syncope, or hospital admission with receipt of an urgent computed tomography scan of the head.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Garg, Principal Investigator — London Health Sciences Centre Research Institute
Locations (1):
- London Health Sciences Centre Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The dataset from this study is held securely in coded form at ICES. While legal data sharing agreements between ICES and data providers (e.g., healthcare organizations and government) prohibit ICES from making the dataset publicly available, access may be granted to those who meet pre-specified criteria for confidential access, available at www.ices.on.ca/DAS (email: das@ices.on.ca). The full dataset creation plan and underlying analytic code are available from the authors upon request, understanding that the computer programs may rely upon coding templates or macros that are unique to ICES and are therefore either inaccessible or may require modification.

REFERENCES:
- [Background] Bathini L, Jeyakumar N, Sontrop J, McArthur E, Kang Y, Luo B, Bello A, Collister D, Ahmed S, Kaul P, Youngson E, Braam B, Melamed N, Hladunewich M, Garg AX. Impact of Baseline Kidney Function on the Rate of Progressive Kidney Disease After Pregnancy: A Population-Based Cohort Study Research Protocol. Can J Kidney Health Dis. 2025 Feb 28;12:20543581251318836. doi: 10.1177/20543581251318836. eCollection 2025. PMID 40027936
- [Background] Shu D, Zou G, Hou L, Petrone AB, Maro JC, Fireman BH, Toh S, Connolly JG. A simple Cox approach to estimating risk ratios without sharing individual-level data in multisite studies. Am J Epidemiol. 2025 Jan 8;194(1):226-232. doi: 10.1093/aje/kwae188. PMID 38973755
- [Background] Abdullah SS, Rostamzadeh N, Muanda FT, McArthur E, Weir MA, Sontrop JM, Kim RB, Kamran S, Garg AX. High-Throughput Computing to Automate Population-Based Studies to Detect the 30-Day Risk of Adverse Outcomes After New Outpatient Medication Use in Older Adults with Chronic Kidney Disease: A Clinical Research Protocol. Can J Kidney Health Dis. 2024 Jan 6;11:20543581231221891. doi: 10.1177/20543581231221891. eCollection 2024. PMID 38186562
- [Background] Koiso K, Akaza H, Kikuchi K, Aoyagi K, Ohba S, Miyazaki M, Ito M, Sueyoshi T, Matsushima H, Kamimura H, Watanabe T, Higuchi S. Pharmacokinetics of tamsulosin hydrochloride in patients with renal impairment: effects of alpha 1-acid glycoprotein. J Clin Pharmacol. 1996 Nov;36(11):1029-38. doi: 10.1177/009127009603601107. PMID 8973992